CLINICAL TRIAL: NCT06505447
Title: A Three-phase Pilot Study of the Feasibility of the Measurement and Promotion of Sleep and the Circadian Rhythm in a Pediatric Intensive Care Unit
Brief Title: PICU-related Sleep and Circadian Dysregulation Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Amanda B. Hassinger, Clinical Associate Professor of Pediatric Sleep Medicine, State University of New York at Buffalo
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: STUDY ID#00008586
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Circadian Dysrhythmia; Sleep Disturbance; Critical Illness; Children, Only
Keywords: Sleep disruption; circadian rhythm; critical care; pediatrics
MeSH Terms: conditions — Parasomnias; Critical Illness | interventions — Phototherapy

STUDY DESIGN:
Intervention Model Description: Three phase single center pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 1: standard of care (No Intervention): 10 children will be enrolled in the first phase related to determining if using actigraphy and timed saliva melatonin samples can be a feasible way to measure the sleep and circadian rhythm of critically ill children aged 3 to 6 years old while they receive routine critical care.
- Phase 2: Daytime light exposure (Experimental): 10 children will undergo the same sleep monitoring and salivary melatonin sampling as phase 1 while receiving timed exposure to a light box of 10,000 lux within 3 feet of their hospital bed for PICU days #2, 3 and 4.
  Interventions: Other: Daytime light exposure
- Phase 3: Daytime restricted feeding (Experimental): 10 children will undergo the same sleep monitoring and salivary melatonin sampling as phase 1 while attempting to limit all nutrition (parental or enteral) to being provided during the normal hours that the child is awake at home on PICU days #2, 3, 4.
  Interventions: Other: Daytime restricted feeding

INTERVENTIONS:
Other: Daytime light exposure — Participants will be exposed to a 10,000 lux light source within 3 feet of their face/eyes to promote the natural circadian rhythm for 2-3 hours from 10am to 12/1pm depending on their nap time at home
  Other Names: Light therapy
  Arms: Phase 2: Daytime light exposure
Other: Daytime restricted feeding — Participant's nutrition, parenteral or enteral, will be restricted to the hours when they are normally awake at home.
  Arms: Phase 3: Daytime restricted feeding

SUMMARY:
A single center pilot trial investigating the feasibility of using actigraphy and salivary melatonin levels to measure the sleep and circadian rhythm of critically ill children aged 3 to 6 years old. This study will also measure the feasibility of providing daytime light exposure as well as restricting all provided nutrition to during daytime hours.

DETAILED DESCRIPTION:
Several of the identified sleep disruptors in a pediatric intensive care environment may not be modifiable, including restricting feeding to daytime hours and providing normal daytime light exposure. This study aims to measure the feasibility of measuring sleep and circadian patterns in a PICU during routine care and during 2 focused sleep promotion interventions: timed daytime light exposure (DLE) and daytime feeding restriction (DFR). The overall objective of this study is to test the hypothesis that, with multi-disciplinary efforts, providing chronotherapeutic care will be feasible and that reliably measuring sleep patterns and the CR of critically ill children with timed salivary melatonin assays and actigraphy is possible.

ELIGIBILITY:
Inclusion Criteria:

1. Child age 3 to 6 years old on the day of PICU admission
2. English-speaking parent at the bedside
3. Child expected to remain in the PICU over 24 to 48 hours

Exclusion Criteria:

1. Child is in end-of-life care
2. The child is receiving neuromuscular blockade for any reason
3. Caregiver or parent not at the bedside

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of monitoring the sleep and circadian rhythm of critically ill children | PICU Day 1 through 4
  The number of days that reliable sleep and CR data are obtained using an actigraph and serial salivary melatonin assays

SECONDARY OUTCOMES:
Feasibility of providing daytime light exposure | PICU Day 2 through 4
  Feasibility will be defined by the percentage of days when DLE was implemented and the average hours of DLE provided using a bedside DLE log
Feasibility of restricting nutrition to daytime hours | PICU Day 2 through 4
  . The feasibility of daytime restricted feeding will be determined by the percentage of enteral or parenteral nutrition that was provided on each study day outside of the child's daytime feeding period determined by the Intake and Output records in the EMR

CONTACTS AND LOCATIONS:
Locations (1):
- John R. Oishei Children's Hospital, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
Our institution has no current ability to create de-identified data sets available to share at this time, but this could change by study completion.

REFERENCES:
- [Background] Traube C, Silver G, Gerber LM, Kaur S, Mauer EA, Kerson A, Joyce C, Greenwald BM. Delirium and Mortality in Critically Ill Children: Epidemiology and Outcomes of Pediatric Delirium. Crit Care Med. 2017 May;45(5):891-898. doi: 10.1097/CCM.0000000000002324. PMID 28288026
- [Background] Kamdar BB, Kamdar BB, Needham DM. Bundling sleep promotion with delirium prevention: ready for prime time? Anaesthesia. 2014 Jun;69(6):527-31. doi: 10.1111/anae.12686. No abstract available. PMID 24813131
- [Background] Kudchadkar SR, Aljohani OA, Punjabi NM. Sleep of critically ill children in the pediatric intensive care unit: a systematic review. Sleep Med Rev. 2014 Apr;18(2):103-10. doi: 10.1016/j.smrv.2013.02.002. Epub 2013 May 21. PMID 23702219
- [Background] Pun BT, Balas MC, Barnes-Daly MA, Thompson JL, Aldrich JM, Barr J, Byrum D, Carson SS, Devlin JW, Engel HJ, Esbrook CL, Hargett KD, Harmon L, Hielsberg C, Jackson JC, Kelly TL, Kumar V, Millner L, Morse A, Perme CS, Posa PJ, Puntillo KA, Schweickert WD, Stollings JL, Tan A, D'Agostino McGowan L, Ely EW. Caring for Critically Ill Patients with the ABCDEF Bundle: Results of the ICU Liberation Collaborative in Over 15,000 Adults. Crit Care Med. 2019 Jan;47(1):3-14. doi: 10.1097/CCM.0000000000003482. PMID 30339549
- [Background] Berger J, Zaidi M, Halferty I, Kudchadkar SR. Sleep in the Hospitalized Child: A Contemporary Review. Chest. 2021 Sep;160(3):1064-1074. doi: 10.1016/j.chest.2021.04.024. Epub 2021 Apr 22. PMID 33895129
- [Background] Hassinger AB, Mody K, Gomez R, Wrotniak BH, Falkowski K, Breuer R, Mennie C, Flagg LK. Validation of the Survey of Sleep Quality in the Pediatric Intensive Care Unit (SSqPICU). J Clin Sleep Med. 2024 Aug 1;20(8):1251-1258. doi: 10.5664/jcsm.11116. PMID 38456806